CLINICAL TRIAL: NCT03153176
Title: "Escola em Ação": School Based Interventions of Incentive to the Practice Physical and Life Habits of Healthy Promotion
Brief Title: "Escola em Ação" (School in Action)
Acronym: EA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Sueyla Ferreira da Silva dos Santos, Principal Investigator, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UNESP Presidente Prudente
Record Dates: First submitted 2017-05-07; First posted 2017-05-15 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Physical Activity; Eating Behavior; Sedentary Lifestyle; Adolescent Behavior
Keywords: physical activity; physical fitness; eating habits; sedentary behavior; sleep quality; satisfaction personal; school health; adolescent
MeSH Terms: conditions — Motor Activity; Feeding Behavior; Sedentary Behavior; Adolescent Behavior; Sleep Initiation and Maintenance Disorders; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: physical activity and lifestyle intervention
Who Masked: Investigator, Outcomes Assessor
Masking Description: Allocation, and those who evaluate the outcomes of the main outcome (physical activity, sedentary behavior, dietary intake and body composition) will be blind to baseline group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): Training program for Physical Education teacher. Individual level: moderate to vigorous physical activity. Organizational level: school health policy for healthy lifestyle
  Interventions: Behavioral: Training; Behavioral: Individual level; Behavioral: Organizational level
- no intervention (No Intervention): Physical Education and school curriculum as usual

INTERVENTIONS:
Behavioral: Training — Training program 30 hours accumulated before, during and after intervention
  Other Names: Training program for Physical Education teacher
  Arms: intervention
Behavioral: Individual level — 7 to 10 minutes in Physical Education in class time, 3 sections for week during lunch break
  Other Names: Moderate to vigorous physical activity
  Arms: intervention
Behavioral: Organizational level — Inclusion of actions in the school curriculum: counseling sections with health for parents and adolescent, active lesson breaks during theoretical class, gardening experience in school, nutrition guidance for school lunch professionals.
  Other Names: School health policy for healthy lifestyle
  Arms: intervention

SUMMARY:
Background: The health promotion actions carried out in the school environment have positive effects on reducing risk factors for chronic diseases in adolescents. Interdisciplinary strategies involving school and family to increase the level of physical activity among adolescents, inside and outside the school, are essential to encourage healthier lifestyles.

Aim: To determine whether a 24-weeks interdisciplinary intervention program promotes improvement in the level of physical activity, physical fitness, sleep quality, life satisfaction, eating habits and reduce the sedentary behavior of schoolchildren aged 10 to 13 years of public schools in the city of Presidente Prudente, São Paulo, Brazil.

The intervention: Includes training of teacher Physical Education in the principles of self-determination theory and ecological theory at practical applications for motivating adolescents in physical activities and sports. The students will be given information on the benefits of a physically active lifestyle and will be encouraged to participated the new opportunities for physical activity in their school and community. The program will offer physical activity strategies over the 24-weeks during class Physical Education, afternoon recess and active lesson breaks in theoretical classes. Nutritional guidelines and gardening experience will be developed to encourage healthy eating habits among schoolchildren and to reduce salt, oil and sugar in the preparation of school lunch.

Methods/design: The project, which being conducted as cluster randomized trial, is to evaluated whit in a mixed methods, including qualitative and quantitative approach will be used for the construction of the actions integrated to the school physical education curriculum and evaluation of the program by the participants and supporters. The RE-AIM evaluation metric (Reach, Effectiveness, Adoption, Implementation, and Maintenance) is used to guide the validation this program.

DETAILED DESCRIPTION:
The intervention will be unfold over the 24-weeks with students of six to seven school terms of implementation physical activity and nutrition intervention strategies. The total of five schools full-time were contacted for participation in the survey, one was excluded because they had no interest in participating. Allocation of pairs of schools in the experimental and control groups was done by randomization (draw for the experimental and control groups), and later the schools were informed about their condition in the study (experimental group or control group). The dimensions assessed in the research were defined from the problems and needs pointed out by the school in the initial stage of training and diagnosis of the local reality. The intervention strategies consisted of the following across: promote teacher Physical Education training; develop school actions integrated in the school curriculum; increase pratice of physical activity (in class time and recess); Improve eating habits (nutritional guidence, gardening experience, school lunch); promote healthy lifestyle program during school breaks; provided with physical activity equipment; parent engagement in health education practice.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in 2017, in the 6th and 7th year of Elementary School in the full-time schools participating in the study

Exclusion Criteria:

* Students with physical or motor impairment that prevents the performance of physical fitness assessments or with mental or cognitive impairment that prevents them from responding with clarity to the questionnaires and instruments of data collection

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 357 (Actual)
Dates: Start 2017-05-08 (Actual); Primary Completion 2017-06-09 (Actual); Study Completion 2018-12-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in weekly time in moderate-to-vigorous physical activity at six months | Baseline, end of intervention (6 months), 1 year after baseline
  Measured with accelerometers for tenn days and supplemented with a questionnaire
Change from baseline in weekly time in sedentary activity at six months | Baseline, end of intervention (6 months), 1 year after baseline
  Measured with accelerometers for tenn days and supplemented with a questionnaire

SECONDARY OUTCOMES:
Change from baseline in Physical Education class time in moderate-to-vigorous physical activity at six months | Baseline, end of intervention (6 months), 1 year after baseline
  Measured with accelerometers in Physical Education class
Change from baseline in level physical fitness at six months | Baseline, end of intervention (6 months), 1 year after baseline
  Measured with physical fitness test (abdominal resistance, palmar grip, horizontal jump, Wells bench, beep test)
Change from baseline in body composition at six months | Baseline, end of intervention (6 months), 1 year after baseline
  Measured with Dual-energy X-ray absorptiometry (DXA) and anthropometric measurements (body height, body weight, waist circumference, hip circumference, arm circumference, triceps skin fold and puberty status (self- assessed)
Change from baseline in caloric intake at six months | Baseline, end of intervention (6 months), 1 year after baseline
  Measured with food register at 3 days and supplemented with a questionnaire

OTHER OUTCOMES:
Change from baseline in the time and quality sleep at six months | Baseline, end of intervention (6 months), 1 year after baseline
  Measured with accelerometers for tenn days and supplemented with a questionnaire (Pittsburgh sleep quality index)
Change from baseline in performance academic at six months | Baseline, end of intervention (6 months), 1 year after baseline
  Measured with school scores and state education performance exam
Change from baseline in satisfaction with life at six months | Baseline, end of intervention (6 months), 1 year after baseline
  Measured with standardized questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ismael Freitas Junior, Phd, Study Director — CELAPAM
Locations (1):
- Sueyla Ferreira da Silva dos Santos, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
This sharing is available for principal researchers and collaborators and may be obtained by individual report after data analysis

REFERENCES:
- [Derived] Ferreira da Silva Dos Santos S, Bordin D, Dornelas de Souza EF, Freitas Junior IF. Study protocol and baseline characteristics of "SCHOOL IN ACTION" program on support to physical activity and healthy lifestyles in adolescents. Contemp Clin Trials Commun. 2019 Dec 14;17:100505. doi: 10.1016/j.conctc.2019.100505. eCollection 2020 Mar. PMID 32211554